CLINICAL TRIAL: NCT02370303
Title: A Pilot Study to Isolate and Test Circulating Tumor Cells Using the ClearCell® FX EP+ System
Brief Title: A Study to Isolate and Test Circulating Tumor Cells Using the ClearCell® FX EP+ System
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Clearbridge Biomedics (Industry)
Responsible Party: Principal Investigator, Dennis Wigle, PI, Mayo Clinic
Other Study IDs: 14-003962
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Lung Cancer; Lung Neoplasms; Cancer of Lung; Cancer of the Lung; Neoplasms, Lung; Neoplasms, Pulmonary; Pulmonary Cancer; Pulmonary Neoplasms; Carcinoma, Non-small-cell Lung; Adenocarcinoma; Squamous Cell Carcinoma
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Preoperative blood sample, tumor tissue from lung resection, postoperative blood sample
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to isolate and measure circulating tumor cells in the blood stream to advance detection of cancer and treatment monitoring. In this study, the investigators will utilize the novel technology for circulating tumor cell detection in order to evaluate their presence in patients with lung cancer.

DETAILED DESCRIPTION:
The plan is to collect both blood and tumor samples from the patient's lung cancer in order to validate this technology in detecting circulating tumor cells. The investigators will also obtain a postoperative blood sample to see if there is a decrease in the overall circulating tumor cell measurement once the tumor has been surgically removed.

ELIGIBILITY:
Inclusion Criteria:

* Stage IB and above non-small cell lung cancer or metastatic lung cancer
* Age >18 years old
* Willing and able to consent to study
* No prior history of neoadjuvant therapy.

Exclusion Criteria:

* Age <18 years old
* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a stage IB or above non-small cell lung cancer or metastatic cancer undergoing lung surgery at the Mayo Clinic in Rochester, MN.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2014-08; Primary Completion 2016-07-09 (Actual); Study Completion 2016-07-09 (Actual)

PRIMARY OUTCOMES:
Number and types of mutations in the primary tumor. | Within 1 year
Number and type of mutations detectable in the matched circulating tumor cell samples. | Within 1 year

SECONDARY OUTCOMES:
Concordance of mutations detected by either method. | Within 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Wigle, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States